CLINICAL TRIAL: NCT03218488
Title: An Observational Post-authorization Safety Study of Ustekinumab in the Treatment of Pediatric Patients Aged 6 Years and Older With Moderate to Severe Plaque Psoriasis
Brief Title: A Safety Study of Ustekinumab in the Treatment of Pediatric Participants Aged 6 Years and Older With Moderate to Severe Plaque Psoriasis
Acronym: STELARA
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108277; CNTO1275PSO4056 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants 6-17 years of Age With Moderate to Severe Plaque Psoriasis: All Participants diagnosed with moderate to severe plaque psoriasis who will either start therapy with ustekinumab within 2 months after the first assessment in the study or have started therapy with ustekinumab in the 12-week period before the first assessment in the study as per routine clinical practice, will be monitored for the long-term safety of ustekinumab and long-term effects of ustekinumab on growth and development. The primary data source for the study will be the medical records of participants and standardized questionnaires (completed by the physician and by the participant/parent).
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Participants will not receive any intervention as part of this study. Participants with moderate to severe plaque psoriasis who are initiating treatment with ustekinumab in clinical practice (patients should either start therapy with ustekinumab within 2 months after the first assessment in the study or have started therapy with ustekinumab in the 12-week period before the first assessment in the study for the treatment of psoriasis) will be observed for the long-term safety of ustekinumab and the long-term effects of ustekinumab on growth and development.
  Other Names: STELARA

SUMMARY:
The purpose of this study is to monitor the long-term safety of ustekinumab in pediatric participants (6 years to 17 years of age at the time of inclusion) with moderate to severe plaque psoriasis, through monitoring for the following adverse events potentially related to immune modulation: serious infections, malignancies and autoimmunity; and to monitor the long-term effects of ustekinumab on growth (weight, height, body mass index) and development (sexual maturity based on the Tanner Scale).

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of moderate to severe chronic plaque psoriasis
* Either start therapy with ustekinumab for the treatment of psoriasis within 2 months after the first assessment in the study or have started therapy with ustekinumab in the 12-week period before the first assessment in the study; a. the treatment decision must have been taken independently of and prior to a participant's inclusion in the study; b. where participants have started therapy with ustekinumab before the first assessment in the study, appropriate baseline data at the start of ustekinumab treatment must be documented, including psoriasis area and severity index (PASI), physician global assessment of disease (PGA), body surface area (BSA) and children's dermatology life quality index (CDLQI) scores where available
* Participants (and/or a legally-acceptable representative/guardian where applicable) must sign a participation agreement/informed consent form (ICF) allowing source data collection and verification in accordance with local requirements and the participants (and/or a legally-acceptable representative/guardian where applicable) must be able to understand and complete the requested patient-reported outcomes (PROs)
* Be willing to participate in the study

Exclusion Criteria:

* Is enrolled in an interventional clinical study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of pediatric participants (6 years to 17 years of age at the time of inclusion) with a diagnosis of moderate to severe plaque psoriasis who are initiating treatment with ustekinumab in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2032-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Baseline up to end of data collection ((maximum of 8 years)
  An adverse event is any untoward medical occurrence in a patient administered a medicinal product. An adverse event does not necessarily have a causal relationship with the treatment. An adverse event can be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
  All participants will be monitored for the long-term safety of ustekinumab for the frequency and severity of adverse events potentially related to immune modulation and of clinical interest such as: serious infections, malignancies, and autoimmunity.
Evaluation of Growth: Height | Baseline up to end of data collection (maximum of 8 years)
  Growth will be based on height recorded at baseline and throughout the observational period.
Evaluation of Growth: Weight | Baseline up to end of data collection (maximum of 8 years)
  Growth will be based on body weight recorded at baseline and throughout the observational period.
Evaluation of Growth: Body Mass Index (BMI) | Baseline up to end of data collection (maximum of 8 years)
  Growth will be based on body weight recorded at baseline and throughout the observational period. Sex and age adjusted BMI will be calculated by dividing the body weight (in kilograms) by the square of height (in meters).
Sexual Maturity Based on the Tanner scale | Baseline up to end of data collection (maximum of 8 years)
  The Tanner scale is used to measure visible changes during puberty commonly referred to as "Tanner stages". It has 3 components: breasts/genitalia, pubic hair, and growth. Female participants are evaluated for breast development and pubic hair distribution and male participants are evaluated for development of external genitalia and pubic hair distribution, based on a 5-stage ordinal scale ranging from TS 1 (prepubertal/preadolescent characteristics) to TS 5 (mature or adult characteristics).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 50 Response | Baseline up to end of data collection (maximum of 8 years)
  The PASI is a measure for assessing and grading the severity and extent of psoriatic lesions and their response to therapy. The PASI measure also accounts for body surface area of psoriasis involvement. In the PASI measure, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4. Total PASI score ranges from 0 to 72. A PASI 50 response represents at least 50 percent improvement from baseline in the PASI score.
Percentage of Participants Achieving PASI 75 Response | Baseline up to end of data collection (maximum of 8 years)
  The PASI is a measure for assessing and grading the severity and extent of psoriatic lesions and their response to therapy. The PASI measure also accounts for body surface area of psoriasis involvement. In the PASI measure, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4. Total PASI score ranges from 0 to 72. A PASI 75 response represents at least 75 percent improvement from baseline in the PASI score.
Percentage of Participants Achieving PASI 90 Response | Baseline up to end of data collection (maximum of 8 years)
  The PASI is a measure for assessing and grading the severity and extent of psoriatic lesions and their response to therapy. The PASI measure also accounts for body surface area of psoriasis involvement. In the PASI measure, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4. Total PASI score ranges from 0 to 72. A PASI 90 response represents at least 90 percent improvement from baseline in the PASI score.
Percentage of Participants Achieving a Physician's Global Assessment (PGA) Score of 0 or 1 | Baseline up to end of data collection (maximum of 8 years)
  The PGA documents the physician's assessment of the severity of the participant's psoriasis lesions at a given time on a 5-point scale, where (0) = cleared, (1) = minimal, (2) = mild, (3) = moderate, (4) = marked, and (5) = severe. Overall lesions are graded for induration, erythema, and scaling. The sum of the 3 scores will be divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease.
Percentage of Participant's Body Surface Area (BSA) Covered by Plaque-type Psoriasis | Baseline up to end of data collection (maximum of 8 years)
  Percentage of participant's body surface area covered by plaque-type psoriasis was estimated using the palm method: the area equivalent to the participant's palm extending to the proximal interphalangeal joints and thumb = 1 percent (%) of BSA. The total BSA affected was the summation of the BSA of the individual regions affected.
Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) | Baseline up to end of data collection (maximum of 8 years)
  The Children's Dermatology Quality Life Index (CDLQI) questionnaire is used to assess the participant's perspective on the impact of skin disorders on daily living. It is a 10 item instrument with 4-item response options on a scale from 0 (Not at all) to 3 (Very much) and a recall period of 1 week. The total score ranges from 0 to 30, with lower scores indicating better quality of life.
Number of Participants With Comorbidities | Baseline up to end of data collection (maximum of 8 years)
  Participants are assessed for pre-existing and new comorbidities associated with pediatric plaque psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (30):
- Uniklinik Graz, Graz, Austria
- Belgium (4):
  - UCL Hopital Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
  - Grand Hôpital de Charleroi, Loverval
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Herlev Hospital, Hellerup
- France (7):
  - CH Victor Dupouy Argenteuil, Argenteuil
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Groupe Hospitalier Pellegrin CHU de Bordeaux, Bordeaux
  - ICH Hopital A. Morvan, Brest
  - Le Bateau Blanc, Martigues
  - Hopital Necker Enfants Malades, Paris
  - CHU Saint Etienne Hopital Nord, Saint-Etienne
- Germany (3):
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Gemeinschaftspraxis Dres. Quist, Mainz
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Greece (2):
  - Andreas Sygros Hospital, Athens
  - University Hospital for Skin and Venereal Diseases, Thessaloniki
- Radboudumc, Nijmegen, Netherlands
- Oslo universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Russia (4):
  - Moscow Research-Practical Center of Dermatovenerology and Cosmetology, Moscow
  - FSBI 'Scientific Centre of Children Health' of the Russian Academy of Medical Sciences, Moscow
  - Llc Ultramed, Omsk
  - Saint-Petersburg State Pediatric Medical Academy of RosZdrav, Saint Petersburg
- Kinderspital Zürich, Zurich, Switzerland
- United Kingdom (4):
  - University Hospital of Wales, Cardiff
  - Whipps Cross University Hospital, London
  - Great Ormond Street Hospital, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency